CLINICAL TRIAL: NCT02495103
Title: Phase I/II Trial of Vandetanib in Combination With Metformin in Subjects With HLRCC or SDH-Associated Kidney Cancer or Sporadic Papillary Renal Cell Carcinoma
Brief Title: Vandetanib in Combination With Metformin in People With HLRCC or SDH-Associated Kidney Cancer or Sporadic Papillary Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Vandetanib is no longer available as Sanofi has decided not to provide additional drug. All subjects are off-study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ramaprasad Srinivasan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150157; 15-C-0157
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Renal Cell Carcinoma; Hereditary Leiomyomatosis; Renal Cell Cancer
Keywords: Dose-Escalation; Maximum Tolerated Dose; Overall Response
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — vandetanib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I Component - Vandetanib (Experimental): Phase I Component
  Interventions: Drug: Vandetanib; Drug: Metformin
- Phase II Component- Vandetanib/Metformin (Experimental): Phase II Component
  Interventions: Drug: Vandetanib/Metformin

INTERVENTIONS:
Drug: Vandetanib — PHASE I: Vandetanib by mouth (PO) daily at 300mg in combination with escalating doses of metformin.
  Other Names: Caprelsa
  Arms: Phase I Component - Vandetanib
Drug: Metformin — Phase I: Metformin starting dose 250mg by mouth (PO) daily in combination with Vandetanib
  Other Names: Glucophage
  Arms: Phase I Component - Vandetanib
Drug: Vandetanib/Metformin — Phase II: Vandetanib and metformin by mouth (PO) daily at determined maximum tolerated dose (MTD).
  Arms: Phase II Component- Vandetanib/Metformin

SUMMARY:
Background:

- There are no established treatments for people with certain advanced kidney cancers. These tumors often don't respond well to currently available treatments. Researchers believe that two drugs that treat other diseases metformin and vandetanib could help people with advanced kidney cancer.

Objective:

- To test the combination of metformin and vandetanib in people with advanced kidney cancer. Phase I of the study will determine a safe dose for the drugs. Phase II will test this dose in people with certain kidney cancers.

Eligibility:

* For Phase I, people 18 and over with advanced kidney cancer
* For Phase II, people 18 and over with advanced hereditary leiomyomatosis and renal cell cancer (HLRCC), succinate dehydrogenase renal cell carcinoma (SDH-RCC), or advanced papillary renal cell carcinoma not related to a hereditary syndrome

Design:

* The study will last many months.
* Participants will be screened with medical history and physical exam.
* Participants will take the study drugs by mouth every day.
* Participants will measure and record their blood pressure every day.
* Participants will have many tests:
* Blood and urine tests
* Magnetic resonance imaging (MRI), computed tomography (CT), positron emission tomography (PET) scan, and other imaging tests: they will lie in machines that take pictures of their body.
* Electrocardiogram (ECG): soft electrodes will be stuck to the skin. A machine will record the hearts signals.
* Bone scan
* Some participants may have a gynecology evaluation or photos of skin tumors taken.
* Participants will have an optional tumor biopsy.
* After they stop taking the drugs, participants may have medical history, physical exam, and blood tests. They will be contacted once a year by phone to find out how they are doing.

DETAILED DESCRIPTION:
BACKGROUND:

* The management of advanced renal cell carcinoma (RCC) continues to remain a challenge, particularly for patients with papillary and non-clear cell variants of RCC, for whom there is no standard therapy of proven benefit.
* Inactivation of the Krebs cycle enzyme Fumarate Hydratase (FH) in tumors associated with hereditary leiomyomatosis and renal cell cancer (HLRCC) results in a metabolic shift characterized by a) reliance on aerobic glycolysis for energy production, b) upregulation of hypoxia-inducible factor 1 (HIF 1-) and its downstream targets that promote glucose delivery and uptake to fuel aerobic glycolysis, and c) downregulation of 5' AMP-activated protein kinase (AMPK), resulting in activation of the mammalian target of rapamycin (mTOR) pathway and increased macromolecule synthesis.
* Inactivation of another Krebs cycle enzyme, Succinate Dehydrogenase (SDH), is also associated with a familial form of kidney cancer which shares some of the above metabolic features.
* Vandetanib is a dual Vascular endothelial growth-factor receptor (VEGFR)/estimated glomerular filtration rate (EGFR) inhibitor that reverses the metabolic phenotype associated with fumarate hydratase (FH) (and SDH) inactivation and has potent preclinical activity in FH-/- and SDH -/- tumors. Metformin activates AMPK and has demonstrated potent synergy when combined with vandetanib, in preclinical models of FH -/- tumors.
* In this phase 1/2 trial, we first propose to establish the safety and dosing parameters of combined vandetanib and metformin therapy. We then propose to test the activity of vandetanib in combination with metformin in patients with HLRCC or SDH-associated RCC, as well as those with sporadic forms of papillary RCC.

OBJECTIVE:

Phase I Component:

-Establish the safety and maximum tolerated dose of the combination of vandetanib with metformin in patients with advanced RCC.

Phase II Component:

-Determine the overall response rate (Response Evaluation Criteria in Solid Tumors (RECIST 1.1) following treatment with combine vandetanib/metformin in patients with 1) advanced RCC associated with hereditary leiomyomatosis and renal cell carcinoma (HLRCC) or succinate dehydrogenase renal cell carcinoma (SDH-RCC), and 2) advanced sporadic papillary renal cell carcinoma.

ELIGIBILITY:

Phase I Component:

* Diagnosis of advanced RCC
* Patients with clear cell RCC must have either declined, be unable to receive, progressed on, or be intolerant of high-dose IL-2 or established first and second line VEGF and/or mTOR targeted agents
* No prior therapy is required in patients with non-clear cell RCC, but prior therapy is allowed

Phase II Component:

* Diagnosis of advanced RCC associated with HLRCC or SDH-RCC (cohort 1) or sporadic/non-HLRCC papillary RCC (cohort 2)
* No more than 2 prior regimens with VEGF-pathway antagonists

General requirements for both Phase I and II:

* Age greater than or equal to18
* Brain metastases or spinal cord compression that requires treatment, unless the treatment ended at least 4 weeks before starting protocol therapy and the condition has been stable without steroid treatment for at least 10 days
* No major surgery within four weeks or inadequately healed wounds prior to study enrollment
* Adequate organ function

DESIGN:

Phase I Component:

* Combination vandetanib and metformin will be administered at starting doses of 300 mg every day (QD) and 250 mg twice a day (BID), respectively.
* The study design is based on a single arm, fixed order dose-escalation Phase 1 study using a modified Fibronacci schema.
* Up to 6 patients may be enrolled in a specific dose combination cohort. Based on the assumption that 3 dose levels will be evaluated, the total number of evaluable patients will be 18. To allow for a few patients who may be inevaluable, the accrual ceiling for this portion of the study will be set at 21. Based on how dose escalation proceeds and the adverse events seen, the total number of patients to be accrued may be changed via a protocol amendment.

Phase II Component:

* Once the maximum tolerated dose (MTD) is determined, the appropriate combination dose will be evaluated in the phase 2 component.
* Patients will be accrued into one of two independent, parallel cohorts:

  * Cohort 1 Patients with advanced HLRCC or SDH associated RCC.
  * Cohort 2 Patients with advanced sporadic/non-HLRCC papillary kidney cancer.
* Patients will be evaluated for response every 8-12 weeks using RECIST 1.1.
* The study is based on open label two-stage optimal phase II design.
* The accrual ceiling for this portion of the study will be 21 patients for each cohort.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis/Histology

     1. Phase I Component - Histologically confirmed advanced Renal Cell Carcinoma (RCC) of any subtype.
     2. Phase II Component - Advanced RCC associated with 1) Hereditary leiomyomatosis and renal cell carcinoma (HLRCC) or Succinate dehydrogenase (SDH) (Cohort 1); OR 2) advanced non HLRCC-related papillary RCC (Cohort 2).
  2. Phase 1: Patients must have evaluable disease

Phase 2: Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan or magnetic resonance imaging (MRI) (except for lymph nodes, which must be >15 mm).

3. Prior Therapy

1. Phase 1- Patients with clear cell RCC must have either declined, be ineligible to receive, have progressed on, or be intolerant to high dose Interleukin 2 (IL-2), or standard first and second line Vascular endothelial growth factor (VEGF), or mammalian target of rapamycin (mTOR) targeted agents. As there is no standard therapy for metastatic non-clear cell RCC, no prior therapy is required.
2. Phase 2- No more than two prior VEGF-pathway targeted agents
3. No previous treatment with vandetanib. Previous or ongoing treatment with metformin is allowed.

   4. Age greater than or equal to18 years.

   5. Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%).

   6. Negative pregnancy test (urine or serum) for female patients of childbearing potential.

   7. Patients must have normal organ and marrow function as defined below:

   absolute neutrophil count greater than or equal to 1,500/mcL

   platelets greater than or equal to 100,000/mcL

   total bilirubin less than or equal to 1.5x upper limit of reference range ( < 3x upper limit of reference range in patients with Gilbert's disease)

   aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)(Serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 X institutional upper limit of normal

   Estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) greater than or equal to 50 mL/min/1.73 m^2

   8. Men and women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for at least 6 months after vandetanib/metformin therapy. Should a woman become pregnant (either a participant or the partner of a male participant) or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

   9. Ability of subject to understand and the willingness to sign a written informed consent document.

   EXCLUSION CRITERIA:
   1. Known serious allergic reaction to vandetanib or metformin.
   2. Brain metastases or spinal cord compression that requires treatment, unless the treatment ended at least 4 weeks before starting protocol therapy and the condition has been stable without steroid treatment for at least 10 days.
   3. Major surgery (includes any surgery that carries significant risk of blood loss, extended periods of general anesthesia, or requires at least an overnight hospital admission) within 28 days before starting treatment or inadequately healed incision/scar from prior surgery.
   4. Any unresolved chronic toxicity greater than Common Terminology Criteria for Adverse Event (CTCAE) Grade 2 or greater from previous anti-cancer therapy (this criterion does not apply to alopecia).
   5. Unacceptable electrolyte values, including:

      * Potassium <4.0 mmol/L despite supplementation, or elevated potassium above the CTCAE Grade 1 upper limit.
      * Magnesium below the lower limit of normal range despite supplementation, or elevated magnesium above the CTCAE Grade 1 upper limit.
      * Ionized calcium or corrected calcium values below the normal range or hypercalcemia above the CTCAE Grade 1 upper limit.
   6. Significant cardiac event (eg, myocardial infarction), New York Heart Association (NYHA) classification of heart disease greater than or equal to 2 within 12 weeks before starting treatment, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
   7. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Patients with atrial fibrillation controlled by medication are permitted.
   8. Hypertension not controlled by medical therapy (systolic blood pressure greater than 140 millimeter of mercury [mmHg] or diastolic blood pressure greater than 90 mmHg).
   9. Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease.
   10. Proteinuria > 1gram/24 hrs
   11. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigators opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
   12. Previous or current invasive malignancies of other histologies requiring treatment within the last 2 years, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin (phase 2 only).

   13 Congenital long Q wave T wave (QT) syndrome.

   14 Any concomitant medications that are known to be associated with Torsades de Pointes Drugs that in the investigators opinion cannot be discontinued, are allowed however, must be monitored closely

   15 .Any concomitant potent inducers of cytochrome P450 3A4 (CYP3A4) function (see http://medicine.iupui.edu/clinpharm/ddis/table.aspx for a continually updated list of CYP3A4 inducers).

   16 History of QT prolongation associated with other medications that required discontinuation of that medication.

   17 Fridericia's (QTcF) correction unmeasurable or >450 ms on screening electrocardiogram (ECG) (Note: If a patient has a QTcF interval >450 ms on screening ECG, the screening ECG may be repeated twice [at least 24 hours apart] for a total of 3 ECGs. The average QTcF from the three

   screening ECGs must be less than or equal to 450 ms in order for the patient to be eligible for the study).

   18. Women that are currently breast feeding.

   19. Active treatment-refractory diarrhea that may affect the ability of the patient to absorb the trial agents or tolerate further diarrhea.

   20. Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with vandetanib/metformin.

   21. Patients with active hemoptysis, clinically significant non hemorrhoidal gastrointestinal (GI) bleeding or those with bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0157.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily: Phase I Component
  Vandetanib: PHASE I: Vandetanib by mouth (PO) daily at 300mg in combination with escalating doses of metformin.
  Metformin: Phase I: Metformin starting dose 250mg by mouth (PO) daily in combination with Vandetanib
- Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily: Phase I Component
  Vandetanib: PHASE I: Vandetanib by mouth (PO) daily at 300mg in combination with escalating doses of metformin.
  Metformin: Phase I: Metformin starting dose 250mg by mouth (PO) twice daily in combination with Vandetanib
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (4.77) | 57.9 (3.07) | 52.03 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Component - Maximum Tolerated Dose (MTD) of Vandetanib and Metformin When Used in Combination in Patients With Metastatic Renal Cell Carcinoma (RCC)
Description: MTD is the dose level at which no more than 1 of up to 6 patients experience dose limiting toxicity (DLT) during 1 cycle of treatment (42 days from the time the intended dose of metformin is reached for a given dose level), and the dose below that at which at least 2 (of ≤6) patients have DLT as a result of the experimental regimen. A DLT is defined as grade III or greater diarrhea leading to hospitalization or lasting > 48 hours despite optimal anti-diarrheal medication; grade IV diarrhea despite optimal anti-diarrheal prophylaxis; grade III or greater nausea or vomiting despite optimal antiemetics; grade III hypertension that is not controlled (to 140/90 mmHg or below) despite optimal antihypertensive therapy; grade III elevated serum creatinine that cannot be corrected to grade 1 or better with hydration within 48 hours; and electrolyte abnormalities that cannot be corrected with medical management within 72 hours.
Time Frame: 42 days after the last patient starts therapy.
Measure: Number; unit: mg
Groups:
- All Participants: All participants that received Phase I, Dose Level 1 - Metformin 250mg daily/Vandetanib 300mg daily; and Phase I, Dose Level 2 - Metformin 250mg twice daily/Vandetanib 300mg daily.
Arm/Group | All Participants
Number analyzed (Participants) | 7
mg | NA — MTD was not reached because accrual was halted before sufficient number of patients could be enrolled for adequate MTD.

2. Primary Outcome: Phase 2 Component - Percentage of Participants With an Overall Response Rate Following Treatment With the Combination of Vandetanib and Metformin
Description: Percentage of participants with an overall response rate following treatment with the combination of vandetanib and metformin in patients with 1) advanced Renal Cell Carcinoma (RCC) associated with Hereditary leiomyomatosis and renal cell cancer (HLRCC) or Succinate Dehydrogenase (SDH), and 2) advanced sporadic/non-HLRCC Papillary Renal Cell Carcinoma assessed by the Response Evaluation Criteria in SOlid Tumors (RECIST) v1.1.
Time Frame: Approximately 8 weeks after initiation of therapy, every 8 weeks thereafter for the first 32 weeks, and then every 12 weeks while on treatment
Population: This outcome measure was not done because we did not enter the phase II portion of the study, thus this endpoint was not evaluated. Vandetanib is no longer available as Sanofi has decided not to provide additional drug.
Groups:
- Phase II Component- Vandetanib/Metformin: Phase II Component- Vandetanib/Metformin
Arm/Group | Phase II Component- Vandetanib/Metformin
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 2 Component - Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was assessed by the and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first
Population: as for outcome 2
Arm/Group | Phase II Component- Vandetanib/Metformin
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 2 Component - Time to Progression (TTP)
Description: Time to progression is the time between the first day of treatment to the day of disease progression. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Phase II Component- Vandetanib/Metformin
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Phase 1 Component - Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily
Number analyzed (Participants) | 3 | 4
Participants | 3 | 4

6. Other Pre Specified Outcome: Phase 1 Component - Number of Participants With a Dose Limiting Toxicity (DLT)
Description: A DLT is defined as grade III or greater diarrhea leading to hospitalization or lasting > 48 hours despite optimal anti-diarrheal medication; grade IV diarrhea despite optimal anti-diarrheal prophylaxis; grade III or greater nausea or vomiting despite optimal antiemetics; grade III hypertension that is not controlled (to 140/90 mmHg or below) despite optimal antihypertensive therapy; grade III elevated serum creatinine that cannot be corrected to grade 1 or better with hydration within 48 hours; and electrolyte abnormalities that cannot be corrected with medical management within 72 hours.
Time Frame: Cycle 1 or 42 days from the time the intended dose of metformin is reached for a given dose level
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 24 months.
Arm/Group | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily (N=3) | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily (N=4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 - Metformin 250mg Daily/Vandetanib 300mg Daily (N=3) | Phase I, Dose Level 2 - Metformin 250mg Twice Daily/Vandetanib 300mg Daily (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (7)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (5) | 3 (8)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (7)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 1 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 2 (6) | 3 (6)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (6)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (3) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 4 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (8)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (3) | 3 (3)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 3 (12)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (4) | 4 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 1 (6)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02495103/Prot_SAP_000.pdf
  • Informed Consent Form: Phase I Standard Consent (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02495103/ICF_001.pdf
  • Informed Consent Form: Phase II Standard Consent (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02495103/ICF_002.pdf